CLINICAL TRIAL: NCT04979598
Title: Unravelling Risk Factors for Chronic Dizziness in Patients After an Acute Unilateral Vestibular Deafferentiation Syndrome.
Brief Title: Unravelling Risk Factors for Chronic Dizziness in Patients After an Acute Unilateral Vestibular Deafferentiation.
Acronym: Activation
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Lien Van Laer, Investigator, Universiteit Antwerpen
Other Study IDs: 42186
Record Dates: First submitted 2021-07-06; First posted 2021-07-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Acute Unilateral Vestibular Deafferentiation
Keywords: Vestibular Neuritis; Labyrinthitis; Vestibular Neurectomy; Resection Vestibular Schwannoma; Gentamicin Injection
MeSH Terms: conditions — Vestibular Neuronitis; Labyrinthitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute unilateral vestibular deafferentiation: Patients suffering from acute dizziness due to a unilateral vestibular deafferentiation.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Home exercise program — A home exercise program is provided but this is an observational study. The effect of the exercise program is not under investigation.

SUMMARY:
In many patients with an acute unilateral vestibular deafferentiation (uVD) syndrome symptoms are expected to resolve spontaneously because of central compensation. However, more detailed observations have revealed that 29-66 % of uVD patients develop disabling chronic dizziness lasting >1 year after the acute event. Identifying predictors of chronic dizziness would allow patients at high risk to be targeted with personalized therapies to reduce healthcare costs. Therefore, the main objective of this study is to identify predictors of chronic dizziness after an acute uVD. Despite the consensus on the usefulness of physical therapy, incorporation of physical therapy programs in daily management of patients after acute uVD remains troublesome. Therefore, the first objective is to study the effect of the actual level of physical activity in the acute stage on long term (LT) outcome. Recent data show that LT prognosis is more linked to anxiety and somatization traits than to objective vestibular findings. Therefore, the second objective is to study the effect of activities avoidance behavior on LT outcome. As stated above it is questioned whether objective vestibular findings can predict chronicity. However recently the Perez and Rey(PR) score was developed. Therefore, the third objective is to study the effect of early central vestibular compensation as measured by the PR score on LT outcome. In patients with poor central vestibular compensation the remaining sensory cues will need to compensate for the loss of vestibular information. Patients using a visual compensation strategy can become dependent of stable visual cues. Therefore, the fourth objective is to study the effect of visual motion sensitivity on LT outcome. A 2-year prospective cohort study will be performed to study aforementioned risk factors for chronic dizziness. Up to 200 consecutive patients with an acute uVD will be included. Chronic dizziness is indicated by a score >30 on the Dizziness Handicap Inventory (primary outcome) after 6 months. Possible risk factors will be evaluated by using MOX1-activity loggers (objective 1), the Vestibular Activities Avoidance Inventory (objective 2), video Head Impulse Testing including the Perez & Rey score (objective 3), Subjective Visual Vertical test and Rod & Disc test (objective 4). Measurements will be taken in the acute phase and 4, 10, 26 and 52 weeks after the acute event.

DETAILED DESCRIPTION:
In humans, acute unilateral peripheral vestibular dysfunction, whether by disease, accident, toxicity or iatrogenic, produces the unilateral vestibular deafferentiation (uVD) syndrome. In many patients, it resolves spontaneously and more or less completely because of central compensation. However, more detailed observations have revealed that 29-66% of uVD patients develop disabling chronic dizziness that lasts more than 1 year after the acute event, irrespective of the underlying etiology and regardless of the way the chronic complaints are documented: clinical bedside tests, vestibulo-ocular reflex(VOR) measurements, balance performance or perceived handicap. Although these chronic symptoms are not severe or life-threatening, they generate significant personal and social handicap in patients, leading to frequent consultations in general practice, Ear-Nose-Throat(ENT) and neurology clinics. A recent epidemiologic study revealed a prevalence of 6.5% of peripheral vestibular disorders in 70.315.919 patients in Germany thereby demonstrating its impact on society in a developed country. Identifying predictors of the "acute-to-chronic" dizziness transition would allow patients at high risk for developing chronic dizziness to be targeted with personalized therapies to reduce healthcare costs. In addition, up to 50% of patients with a chronic vestibular syndrome have a risk of developing depression or anxiety disorders. Therefore, the main objective of this study is to identify predictors of chronicity with a focus on investigating the effect of patients' tendency to avoid complaint-triggering movements and the actual level of physical activity on long-term outcomes in patients after acute uVD. Medical treatment in the acute phase is currently focused on symptomatic treatment with antivertiginous drugs (antihistamines) while motivating and helping patients to move as quickly as possible, an essential part of vestibular rehabilitation. There is moderate to strong evidence that vestibular rehabilitation is a safe, effective management for unilateral peripheral vestibular dysfunction, based on a number of high-quality randomized controlled trials. Furthermore, there is moderate evidence that vestibular rehabilitation resolves symptoms and improves functioning in the intermediate term but there is insufficient evidence to discriminate between different forms of vestibular rehabilitation. Based on a clinical practice guideline from the American Physical Therapy Association (Neurology Section),clinicians may offer specific exercise techniques to target identified impairments or functional limitations and may provide supervised vestibular rehabilitation. Despite the consensus on the usefulness of physical therapy, incorporation of physical therapy programs in daily management of patients after acute uVD remains troublesome. Research into health care utilization in patients with dizziness revealed a low number of visits for vestibular disorders were referred to physical therapy in ambulatory care. Moreover, the confrontation with current practice and the review of research protocols that study long-term outcome after an acute uVD show that the approach usually consists of encouraging patients to move a round as much as possible without the supervision of the physical therapist. Early and active vestibular rehabilitation is crucial. However, there are no known studies that investigate the actual physical activity level and/or exercise adherence in home exercise programs in patients with acute uVD. Therefore, our first objective is to study the effect of physical activity/movement volume in the acute stage on long term outcome after an acute uVD. Furthermore, psychological factors such as anxiety, depression and fear of falling have a negative effect on the outcome of vestibular rehabilitation. Indeed, recent data show that long-term prognosis in vestibular neuritis patients is more linked to anxiety and somatization traits than to objective vestibular findings. Pathophysiologic processes seem to include precipitating events that trigger anxiety-related changes in postural strategies with an increased attention to head and body motion and a cocontraction of leg muscles. Fear of movement in response to injury is a concept first introduced in the field of chronic low back pain, where it was shown that fear of inducing or increasing pain could lead to a maladaptive response of restricting movements and activities. In contrast, the confrontation response leads to increased movement and return to activities. This model can be translated to vestibular disorders as avoiding complaint-inducing movements is a known compensation strategy used by patients with an acute uVD. These physical activities are very important to promote compensation and avoiding them can therefore contribute to greater disability. Therefore, the second objective is to study the effect of activities avoidance behavior on long term outcome after an acute uVD. Acute uVD is defined by the patient history, the clinical examination and often characterized by measurable vestibular parameters using three-dimensional video head impulse testing (vHIT), caloric irrigation, sinusoidal harmonious acceleration testing (SHA) and cervical/ocular vestibular-evoked myogenic potentials (c/o VEMP). However, whether these VOR function measurements can predict chronicity is questioned. Recently a new tool (i.e. the Perez and Rey (PR) score) was developed to characterize the state of vestibular compensation of subjects diagnosed with acute uVD of peripheral origin. The PR score is a measure of temporal organization of the refixation saccades that enables to distinguish clearly and objectively between subjects that are in a compensated or uncompensated vestibular situation. However the PR score has never been studied as a prognostic factor of progression to chronicity. Therefore, the third objective is to study the effect of early central vestibular compensation as measured by the PR score on long term outcome after an acute uVD. Accurate perception of gravity is important for spatial orientation, postural balance, and the regulation of gait. Multiple sensory signals contribute to the central processing of this percept, including signals from visual, vestibular and somatosensory systems. Patients after an acute uVD suffer from a deteriorated sense of spatial orientation, leading to balance problems. In uncompensated vestibular patients the remaining sensory cues will need to compensate for the loss of vestibular information. Recently a reweighting of sensory signals with an increase in visual weight of 20-40% was suggested in patients with a bilateral vestibular function loss. This visual compensation strategy can make some patients dependent of stable visual cues which might lead to visual motion sensitivity. Evidence is mounting that visual field dependency is also a factor contributing to visual vertigo in patients with vestibular disorders. Visually induced dizziness or visual vertigo is a specific form of persistent perceptual postural dizziness which is classified as a chronic functional vestibular disorder. Therefore, the fourth objective is to study the effect of visual motion sensitivity on long term outcome after an acute uVD.

ELIGIBILITY:
Inclusion Criteria:

* Acute unilateral vestibular deafferentiation

Exclusion Criteria:

* Central pathologies and bilateral vestibulopathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute unilateral vestibular deafferentiation
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory | 6 months
  Questionnaire concerning impairments due to dizziness: the higher the score, the bigger the perceived handicap due to dizziness.

SECONDARY OUTCOMES:
Perez-and Rey score | Week 1, 4, 10, 26 & 52
  Temporal organisation of corrective saccades
Mox1loggers | Week 1 & 10
  Level of physical activity
Rod&Disc test | Week 10 & 26
  Visual dependency
Anxiety | Week 1, 4, 10, 26 & 52
  Hospital Anxiety and Depression Scale: two subscales (anxiety and depression). A lower score means less chance on an anxiety or depression disorder.
Avoidance behavior | Week 1, 4, 10, 26 & 52
  Vestibular Activities Avoidance Inventory: the higher the score, the bigger the chance that avoidance behavior is present.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Antwerp, Antwerp, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
A registration at the Research Database Antigoon was submitted and approved. In this way a Data Protection Impact Assessment (DPIA) is performed. A Data Management was published on "dmponline.be".

REFERENCES:
- [Background] Alberts BBGT, Selen LPJ, Verhagen WIM, Pennings RJE, Medendorp WP. Bayesian quantification of sensory reweighting in a familial bilateral vestibular disorder (DFNA9). J Neurophysiol. 2018 Mar 1;119(3):1209-1221. doi: 10.1152/jn.00082.2017. Epub 2017 Dec 13. PMID 29357473
- [Background] Batuecas-Caletrio A, Rey-Martinez J, Trinidad-Ruiz G, Matino-Soler E, Cruz-Ruiz SS, Munoz-Herrera A, Perez-Fernandez N. Vestibulo-Ocular Reflex Stabilization after Vestibular Schwannoma Surgery: A Story Told by Saccades. Front Neurol. 2017 Jan 25;8:15. doi: 10.3389/fneur.2017.00015. eCollection 2017. PMID 28179894
- [Background] Bergenius J, Perols O. Vestibular neuritis: a follow-up study. Acta Otolaryngol. 1999;119(8):895-9. doi: 10.1080/00016489950180243. PMID 10728930
- [Background] Bronstein AM, Dieterich M. Long-term clinical outcome in vestibular neuritis. Curr Opin Neurol. 2019 Feb;32(1):174-180. doi: 10.1097/WCO.0000000000000652. PMID 30566414
- [Background] Cousins S, Cutfield NJ, Kaski D, Palla A, Seemungal BM, Golding JF, Staab JP, Bronstein AM. Visual dependency and dizziness after vestibular neuritis. PLoS One. 2014 Sep 18;9(9):e105426. doi: 10.1371/journal.pone.0105426. eCollection 2014. PMID 25233234
- [Background] Cousins S, Kaski D, Cutfield N, Arshad Q, Ahmad H, Gresty MA, Seemungal BM, Golding J, Bronstein AM. Predictors of clinical recovery from vestibular neuritis: a prospective study. Ann Clin Transl Neurol. 2017 Mar 22;4(5):340-346. doi: 10.1002/acn3.386. eCollection 2017 May. PMID 28491901
- [Background] Dieterich M, Staab JP. Functional dizziness: from phobic postural vertigo and chronic subjective dizziness to persistent postural-perceptual dizziness. Curr Opin Neurol. 2017 Feb;30(1):107-113. doi: 10.1097/WCO.0000000000000417. PMID 28002123
- [Background] Eckhardt-Henn A, Breuer P, Thomalske C, Hoffmann SO, Hopf HC. Anxiety disorders and other psychiatric subgroups in patients complaining of dizziness. J Anxiety Disord. 2003;17(4):369-88. doi: 10.1016/s0887-6185(02)00226-8. PMID 12826087
- [Background] Godemann F, Siefert K, Hantschke-Bruggemann M, Neu P, Seidl R, Strohle A. What accounts for vertigo one year after neuritis vestibularis - anxiety or a dysfunctional vestibular organ? J Psychiatr Res. 2005 Sep;39(5):529-34. doi: 10.1016/j.jpsychires.2004.12.006. Epub 2005 Mar 4. PMID 15992562
- [Background] Goto F, Sugaya N, Arai M, Masuda K. Psychiatric disorders in patients with intractable dizziness in the department of otolaryngology. Acta Otolaryngol. 2018 Jul;138(7):646-647. doi: 10.1080/00016489.2018.1429652. Epub 2018 Jan 31. PMID 29385877
- [Background] Goudakos JK, Markou KD, Psillas G, Vital V, Tsaligopoulos M. Corticosteroids and vestibular exercises in vestibular neuritis. Single-blind randomized clinical trial. JAMA Otolaryngol Head Neck Surg. 2014 May;140(5):434-40. doi: 10.1001/jamaoto.2014.48. PMID 24604142
- [Background] Guajardo-Vergara C, Perez-Fernandez N. A New and Faster Method to Assess Vestibular Compensation: A Cross-Sectional Study. Laryngoscope. 2020 Dec;130(12):E911-E917. doi: 10.1002/lary.28505. Epub 2020 Feb 7. PMID 32031691
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Treatment for Vestibular Disorders: How Does Your Physical Therapist Treat Dizziness Related to Vestibular Problems? J Neurol Phys Ther. 2016 Apr;40(2):156. doi: 10.1097/01.NPT.0000481898.55592.6e. No abstract available. PMID 26934418
- [Background] Halmagyi GM, Weber KP, Curthoys IS. Vestibular function after acute vestibular neuritis. Restor Neurol Neurosci. 2010;28(1):37-46. doi: 10.3233/RNN-2010-0533. PMID 20086281
- [Background] Hulse R, Biesdorf A, Hormann K, Stuck B, Erhart M, Hulse M, Wenzel A. Peripheral Vestibular Disorders: An Epidemiologic Survey in 70 Million Individuals. Otol Neurotol. 2019 Jan;40(1):88-95. doi: 10.1097/MAO.0000000000002013. PMID 30289843
- [Background] Kammerlind AS, Ledin TE, Skargren EI, Odkvist LM. Long-term follow-up after acute unilateral vestibular loss and comparison between subjects with and without remaining symptoms. Acta Otolaryngol. 2005 Sep;125(9):946-53. doi: 10.1080/00016480510043477. PMID 16109673
- [Background] Kammerlind AS, Ledin TE, Odkvist LM, Skargren EI. Influence of asymmetry of vestibular caloric response and age on balance and perceived symptoms after acute unilateral vestibular loss. Clin Rehabil. 2006 Feb;20(2):142-8. doi: 10.1191/0269215506cr886oa. PMID 16541934
- [Background] Kammerlind AS, Ledin TE, Odkvist LM, Skargren EI. Recovery after acute unilateral vestibular loss and predictors for remaining symptoms. Am J Otolaryngol. 2011 Sep-Oct;32(5):366-75. doi: 10.1016/j.amjoto.2010.07.008. Epub 2010 Oct 2. PMID 20888071
- [Background] Lacour M, Bernard-Demanze L. Interaction between Vestibular Compensation Mechanisms and Vestibular Rehabilitation Therapy: 10 Recommendations for Optimal Functional Recovery. Front Neurol. 2015 Jan 6;5:285. doi: 10.3389/fneur.2014.00285. eCollection 2014. PMID 25610424
- [Background] Lahmann C, Henningsen P, Brandt T, Strupp M, Jahn K, Dieterich M, Eckhardt-Henn A, Feuerecker R, Dinkel A, Schmid G. Psychiatric comorbidity and psychosocial impairment among patients with vertigo and dizziness. J Neurol Neurosurg Psychiatry. 2015 Mar;86(3):302-8. doi: 10.1136/jnnp-2014-307601. Epub 2014 Jun 24. PMID 24963122
- [Background] Dunlap PM, Khoja SS, Whitney SL, Freburger JK. Assessment of Health Care Utilization for Dizziness in Ambulatory Care Settings in the United States. Otol Neurotol. 2019 Oct;40(9):e918-e924. doi: 10.1097/MAO.0000000000002359. PMID 31498294
- [Background] Mandala M, Nuti D. Long-term follow-up of vestibular neuritis. Ann N Y Acad Sci. 2009 May;1164:427-9. doi: 10.1111/j.1749-6632.2008.03721.x. PMID 19645942
- [Background] McDonnell MN, Hillier SL. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Cochrane Database Syst Rev. 2015 Jan 13;1(1):CD005397. doi: 10.1002/14651858.CD005397.pub4. PMID 25581507
- [Background] Patel M, Arshad Q, Roberts RE, Ahmad H, Bronstein AM. Chronic Symptoms After Vestibular Neuritis and the High-Velocity Vestibulo-Ocular Reflex. Otol Neurotol. 2016 Feb;37(2):179-84. doi: 10.1097/MAO.0000000000000949. PMID 26719963
- [Background] Peluso ET, Quintana MI, Gananca FF. Anxiety and depressive disorders in elderly with chronic dizziness of vestibular origin. Braz J Otorhinolaryngol. 2016 Mar-Apr;82(2):209-14. doi: 10.1016/j.bjorl.2015.04.015. Epub 2015 Oct 9. PMID 26515771
- [Background] Rey-Martinez J, Batuecas-Caletrio A, Matino E, Perez Fernandez N. HITCal: a software tool for analysis of video head impulse test responses. Acta Otolaryngol. 2015 Sep;135(9):886-94. doi: 10.3109/00016489.2015.1035401. Epub 2015 Apr 9. PMID 25857220
- [Background] Staab JP, Eckhardt-Henn A, Horii A, Jacob R, Strupp M, Brandt T, Bronstein A. Diagnostic criteria for persistent postural-perceptual dizziness (PPPD): Consensus document of the committee for the Classification of Vestibular Disorders of the Barany Society. J Vestib Res. 2017;27(4):191-208. doi: 10.3233/VES-170622. PMID 29036855
- [Background] Strupp M, Magnusson M. Acute Unilateral Vestibulopathy. Neurol Clin. 2015 Aug;33(3):669-85, x. doi: 10.1016/j.ncl.2015.04.012. PMID 26231279
- [Background] van Vugt VA, van der Wouden JC, Essery R, Yardley L, Twisk JWR, van der Horst HE, Maarsingh OR. Internet based vestibular rehabilitation with and without physiotherapy support for adults aged 50 and older with a chronic vestibular syndrome in general practice: three armed randomised controlled trial. BMJ. 2019 Nov 5;367:l5922. doi: 10.1136/bmj.l5922. PMID 31690561
- [Background] Whitney SL, Sparto PJ, Furman JM. Vestibular Rehabilitation and Factors That Can Affect Outcome. Semin Neurol. 2020 Feb;40(1):165-172. doi: 10.1055/s-0039-3402062. Epub 2019 Dec 30. PMID 31887754
- [Background] Yardley L, Redfern MS. Psychological factors influencing recovery from balance disorders. J Anxiety Disord. 2001 Jan-Apr;15(1-2):107-19. doi: 10.1016/s0887-6185(00)00045-1. PMID 11388354
- [Derived] Hallemans A, Van der Boon H, Vereeck L, Van Rompaey V, Van Laer L. The Minimal Clinically Important Difference of the 180 degrees Turn Time During the Instrumented Timed up and Go in Unilateral Vestibulopathies. Physiother Res Int. 2025 Apr;30(2):e70053. doi: 10.1002/pri.70053. PMID 40135683